CLINICAL TRIAL: NCT06425055
Title: Vonafexor Fixed Dose-escalation Safety and Proof-of-concept Study in Patients With at Risk of Progression Alport Syndrome
Brief Title: Vonafexor ALPort Syndrome Efficacy & Safety TRIAl-1 (ALPESTRIA-1)
Acronym: ALPESTRIA-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-208
Record Dates: First submitted 2024-05-14; First posted 2024-05-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary

STUDY DESIGN:
Intervention Model Description: Single arm fixed dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm fixed dose escalation (Experimental): This is a single arm fixed dose escalation with three dose levels of vonafexor, all QD.
  Interventions: Drug: Vonafexor

INTERVENTIONS:
Drug: Vonafexor — * One tablet of a low dose of vonafexor QD from Day 1 to Week 4
  * One tablet of a medium dose of vonafexor QD from Week 5 to Week 8
  * One tablet of a high dose of vonafexor QD from Week 9 to Week 24
  Other Names: EYP001a

SUMMARY:
This study is a proof-of-concept trial of vonafexor safety, its effects on kidney function in subjects with at risk of progression Alport syndrome.

DETAILED DESCRIPTION:
This is a multicenter study and several clinical sites and countries will be involved.

This single arm, fixed dose escalation, open-label, non-randomized study will evaluate three dose levels of vonafexor on safety, tolerability and their effect on kidney function and renal biomarkers in 20 patients with AS at risk of progression.

The total duration of study for a participant will be up to 40 weeks and include a screening period, a treatment period of 24 weeks and a follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (also for legal representatives, as applicable in the US for under eighteen patients).
* Has confirmed diagnosis of Alport syndrome: clinical diagnosis (haematuria, family history, hearing loss, ocular change) OR a kidney biopsy showing glomerular basement membrane abnormalities consistent with AS, AND Genetic confirmation of AS.
* Has eGFR between ≥ 30 and < 90 ml/min/1.73m2.
* Has increased albuminuria criteria i.e. UACR ≥ 300 mg/g.
* If on an angiotensin converting enzyme inhibitor (ACEi) and/or angiotensin receptor blocker (ARB), should be on a stable well tolerated treatment during at least the 60 days prior D1.
* If on Sodium-Glucose Transport Protein 2 (SGLT2), should be on stable well tolerated treatment with SGLT2 during at least 60 days prior D1.
* If patient has a history of arterial hypertension, should be on stable anti-hypertensive therapy for at least 60 days prior to D1 and deemed controlled by the investigator at screening and D1.
* Sexually active female subjects of childbearing potential and sexually mature male subjects must use two acceptable effective methods of contraception for the entire duration of the study and for at least 6 weeks after last dose.
* Has negative results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV).
* Is able to understand all study procedures in the informed consent form (ICF) and willing to comply with all aspects of the protocol.

Exclusion Criteria:

* Is an employee of a site, clinical research organization, vendor, or sponsor involved with this study.
* Is pregnant or breastfeeding.
* Has participated in any investigational drug study within 60 days prior to D1.
* Any clinically significant illness within 30 days before D1 or surgical or medical condition (other than Alport syndrome) that could interfere with the subject's study compliance; confound the study results; impact subject safety.
* Any history of active malignancy within the last 1 year before D1.
* Any other condition or circumstance that, in the opinion of the investigator, may make the subject unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the subject's safety and well-being.
* Has a history of an allergic condition that required the prescription of an emergency epinephrine injection (such as the EpiPen® Auto-Injector).
* Any prohibited co-medications within 30 days prior D1.
* Has ALT or AST above near normal (>1.5×ULN) at baseline.
* Are at high risk for atherosclerotic cardiovascular disease (ASCVD) risk, with an LDL-C level > 160 mg/dL (4.15 mmol/L) and subjects at intermediate risk for ASCVD risk, with a LDL-C level > 190 mg/dL (4.91 mmol/L).
* Has moderate or severe hepatic impairment (Child-Pugh score B or C).
* Is taking CYP3A4/5 inhibitors or inducers.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Event (TEAE) | From first dose of treatment until 2 weeks after last dose of treatment, i.e assessed up to 26 weeks
  To assess the safety and tolerability of vonafexor

SECONDARY OUTCOMES:
Change in eGFR | During on-treatment (assessed up to 24 weeks) and off-treatment periods (assessed up to 36 weeks) compared to baseline
  To determine the on with the off-treatment effect of three dose levels of vonafexor on renal function
Vonafexor plasma concentrations | During on-treatment period, assessed up to 24 weeks
  To determine vonafexor plasma concentrations levels

OTHER OUTCOMES:
Change in albuminuria | During on-treatment (assessed up to 24 weeks) and off-treatment periods (assessed up to 36 weeks) compared to baseline
  To determine the effect of vonafexor on and off treatment on exploratory renal biomarkers
Change in proteinuria | During on-treatment (assessed up to 24 weeks) and off-treatment periods (assessed up to 36 weeks) compared to baseline
  To determine the effect of vonafexor on and off treatment on exploratory renal biomarkers
Change in Neutrophil Gelatinase Associated Lipocalin (NGAL) | During on-treatment (assessed up to 24 weeks) and off-treatment periods (assessed up to 36 weeks) compared to baseline
  To determine the effect of vonafexor on and off treatment on exploratory renal biomarkers

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Dr Eric Wallace - University of Alabama, Birmingham, Alabama
  - Dr Anjay Rastogi - UCLA Health, David Geffen School of Medicine, Los Angeles, California
  - Dr Arnold Silva - Boise Kidney & Hypertension, Boise, Idaho
  - Dr Suneel Udani - NANI Research, Hinsdale, Illinois
  - Dr Tingting Li - Washington University, St Louis, Missouri
  - Dr James Simon - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dr Ankit Mehta - Renal Disease Research Institute, Dallas, Texas
- France (3):
  - Pr Claire Rigothier - CHU De Bordeaux, Bordeaux
  - Dr Moglie Le Quintrec - Hopital Lapeyronie, Montpellier
  - Pr. Bertrand Knebelmann - Necker Enfants Malades, Paris
- Spain (3):
  - Fundacio Puigvert, Barcelona
  - Hospital Virgen de la Arrixaca, El Palmar
  - Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline published results might be shared upon request with researchers who provide a methodologically sound proposal and to achieve objectives as set in the approved proposal.
  IPD will be shared deidentified and from 3 months and ending 5 years following article publication.
Supporting Information: Study Protocol, SAP
Time Frame: From 3 months and ending 5 years following article publication.

REFERENCES:
- [Derived] Rheault MN. Treatment Approaches for Alport Syndrome. J Am Soc Nephrol. 2025 Sep 12;37(1):172-9. doi: 10.1681/ASN.0000000897. Online ahead of print. PMID 40938675